# You Are Being Asked to Be in a Research Study

#### What Is a Research Study?

The main purpose of research studies is to gain knowledge. This knowledge may be used to help others. Research studies are not intended to benefit you directly, though some might.

#### Do I Have to Do This?

No. Being in this study is entirely your choice. If you decide to join this study, you can change your mind later on and withdraw from the research study.

Taking part in a study is separate from medical care. The decision to join or not join the research study will not affect your status as a patient.

#### What Is This Document?

This form is an informed consent document. It will describe the study risks, procedures, and any costs to you.

This form is also a HIPAA Authorization document. It will describe how your health information will be used and by whom.

Signing this form indicates you are willing to take part in the study and allow your health information to be used.

#### What Should I Do Next?

- 1. Read this form, or have it read to you.
- 2. Make sure the study doctor or study staff explains the study to you.
- 3. Ask questions (e.g., time commitment, unfamiliar words, specific procedures, etc.)
- 4. If there will be medical treatment, know which parts are research and which are standard care.
- 5. Take time to consider this, and talk about it with your family and friends.



A Cancer Center Designated by

WINSHIP CANCER

# Emory University and Grady Health System Consent to be a Research Subject / HIPAA Authorization

**EMORY** 

<u>Title</u>: Winship 3286-16 /**CA209-461 Biomarker-driven Phase 2 study of Nivolumab in Advanced Metastatic Non-Small Cell Lung Cancer (NSCLC)** 

Principal Investigator: Rathi Pillai, MD

Sponsor: Rathi Pillai, MD

Supporter: Bristol Myers Squibb

#### Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

#### Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### What is the purpose of this study?

The purpose of this study is to study changes in immune cells (T cells and others) in the blood and tissue of patients with advanced non-small cell lung cancer (NSCLC) who take nivolumab, a treatment that activates your immune system to fight your lung cancer. Nivolumab is available as standard of care treatment and does not require you to participate in a clinical trial. By taking part in this study, you will help us be able to understand better how nivolumab works to activate your immune system against your lung cancer. We plan to enroll 35 patients at Emory and Grady.

Version Date: 02/16/2018 IRB Form 04152016

#### What will I be asked to do?

If you decide to enroll in this study, you will be asked to undergo a biopsy if your oncologist thinks it is possible and safe before you start on nivolumab. This biopsy sample will be tested in an immunology lab here at Emory and Grady Health System. You will then start on nivolumab and get treatments (infusions) every two weeks in the clinic. You will have to come in for an extra visit the first week after you start on nivolumab. We will draw some extra tubes of blood from you at each of these visits. This blood will be studied in the lab to be able to look at your T cells and other immune cells more closely and to do genetic testing on these immune cells to understand how the nivolumab is working on your immune system.

You will get scans every 6 weeks to see if the nivolumab treatment is controlling your cancer. You will continue on nivolumab as long as it is helping you and your cancer. You will continue to get scans every 6 weeks up until week 49 and then will only get scans every 12 weeks. If the nivolumab is not controlling your cancer, then your doctor will talk to you about stopping it and if you are willing, to get another biopsy when you stop treatment. This biopsy would be studied to understand why the nivolumab stopped working on your cancer.

Some patients will be asked if they would be willing to get a biopsy while they are on treatment at the second cycle. This is completely optional and will be used to understand how immune cells work inside your tumor when you take nivolumab.

#### Who owns my study information and samples?

If you join this study, you will be donating your samples and study information. You will not receive any compensation if your samples or information are used to make a new product. If you withdraw from the study, data and samples that were already collected may be still be used for this study. However, if you do not want us to use your samples when you withdraw from the study, you can request that we destroy any samples we have already collected on you.

#### What are the possible risks and discomforts?

The biopsy that is obtained before you start on the study and additional biopsies that may be obtained during your treatment could be associated with risks. Your treating doctor will discuss with you the safest tumor that can be sampled for the purpose of the study biopsy. This may involve a CT guided biopsy by a radiologist of a tumor in your lung or in your abdomen (such as the liver or a lymph node). Another method is a biopsy of your lung or lymph nodes by your airway involved with cancer via bronchoscopy by an interventional pulmonologist. The potential risks of this biopsy include bleeding, infection, and pain. In the case of a lung biopsy (either CT-guided or by bronchoscopy), there is a risk of collapse of your lung (pneumothorax). If your lung collapses, you would have to stay in the hospital to be treated with a chest tube to help your lung re-expand.

There may be side effects from the study drug (nivolumab) or procedures that are not known at this time.

The most common risks and discomforts expected in this study from nivolumab are:

- Fatigue
- Skin reactions: including rash, itching, hives, redness, and dry skin. Toxic epidermal
  necrolysis, a potentially life threatening disease characterized by blistering and peeling of the

top layer of skin resembling that of a severe burn, has occurred in one patient who received ipilimumab after nivolumab treatment.

- Diarrhea
- Nausea
- Abdominal pain
- Decreased appetite
- Low red blood cells
- Fever
- Joint pain or stiffness

The less common risks and discomforts expected in this study are:

- Bowel inflammation
- Liver function blood test abnormalities
- · Loss of color (pigment) from areas of skin
- Dry mouth
- Vomiting
- Weight loss
- Thyroid gland abnormalities
- Blood chemistry abnormalities, including low blood phosphate, magnesium, and potassium levels.
- High blood uric acid level
- Lung inflammation (pneumonitis see details below)
- Cough
- Dizziness
- Headache
- Low white blood cells
- Chills
- Muscle soreness, weakness, stiffness spasms or paralysis
- Pain in arms or legs
- Tingling, burning, or numbness in hands and feet
- Shortness of breath
- Abnormal taste
- Flushing
- High or low blood pressure
- Allergic reaction during or between study drug infusions
- Increased sensitivity of skin to sunlight
- Constipation
- Difficulty swallowing
- Heartburn
- Low blood platelets (may increase risk of bleeding)

#### Rare but possible risks include:

- Low blood oxygen level
- Acute lung injury or failure
- Collection of fluid around the lungs

Version Date: 02/16/2018 IRB Form 04152016

- Inflammation of the appendix
- Increase in inflammatory blood proteins (e.g., lipase)
- Adrenal gland abnormalities
- Pituitary gland inflammation
- Changes in vision (including decreased or blurry vision), inflammation of the eye, or bleeding into the eye
- Liver inflammation
- Acute kidney injury or failure
- Abnormal blood cell production
- Inflammation of the mouth and lining of the digestive tract
- Swelling of the face, arms, or legs
- Inflammation of the pancreas
- Back pain
- Autoimmune disorders, including Guillain-Barre syndrome (associated with progressive muscle weakness or paralysis)
- Chest discomfort
- Heart palpitations
- Inflammation of the heart or its lining
- Collection of fluid around the heart
- Increased blood sugar
- Dehydration
- Infections: including sepsis, lung infections, and skin infections.
- Decreased movement of the intestines
- Disorientation
- Swelling of the optic disc
- Inflammation of the optic nerve
- Inflammation or loss of the lining of the brain and spinal cord
- Drug reaction with rash, blood cell abnormalities, enlarged lymph nodes, and internal organ involvement (including liver, kidney, and lung); known as Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS)
- Myasthenia gravis, a nerve disease that may cause weakness of eye, face, breathing, and swallowing muscles. One death in a patient who received nivolumab combined with ipilimumab was considered due to myasthenia gravis and severe infection (sepsis).
- Abnormal brain function due to brain inflammation.
- Rhabdomyolysis (muscle fiber released into the blood stream which could damage your kidney) and polymyositis (chronic muscle inflammation with muscle weakness) has been reported in one patient.
- Lung Inflammation (pneumonitis): It is possible that nivolumab may cause inflammation of the tissues of the lung. This adverse effect has been reported infrequently in patients treated with nivolumab. While many patients with x-ray or CT abnormalities have not developed any symptoms, some patients have developed mild to severe symptoms and in rare cases, death has occurred as a result of their lung inflammation. Signs and symptoms of lung inflammation may include difficulty breathing, pain or discomfort while breathing, chest pain, cough, shortness of breath, increased rate of breathing, fever, low blood oxygen levels, or fatigue.

Version Date: 02/16/2018 IRB Form 04152016 Study No.: CA209-461

Your study doctor and nurse will watch you closely for changes in your ability to breathe and for other signs or symptoms that might show you are developing this type of lung inflammation and will perform regular tests including physical exams, measurement of oxygen levels through non-invasive testing (i.e., pulse oximeter), blood tests, chest x-rays and/or CT scans.

# Please inform your study doctor or nurse <u>AT ONCE</u> if you experience any of the following:

- Any new or increased shortness of breath;
- Any new or increased chest pain;
- Any new or increased pain/difficulty while breathing;
- Any new or increased cough or any significant change in your type of cough; for example any new or increased mucous or blood in your cough;
- Any change in the amount of oxygen you require;
- Any fever, fatigue, or other symptoms that occur at the same time as any changes to your breathing or other lung symptoms.

If you start to develop symptoms, your study doctor will ask you to return to the clinic for additional tests, which could include a physical exam, measurement of oxygen levels, blood tests, chest x-rays, and/or CT scans. You will be monitored very closely for changes in your overall lung symptoms, monitoring may require hospitalization. You may require specific treatment in order to control pneumonitis. A special doctor called a pulmonologist, who has special training to be an expert in how your lungs work, may also see you.

Prolonged treatment with medicines that suppress inflammation, sometimes needed to manage the side effects of nivolumab treatment, may lower your body's ability to fight off certain infections (i.e., opportunistic infections). These infections may require treatment with antibiotic or antifungal medications and may be fatal.

If you are a woman: to protect against possible side effects of the study drug, women who are pregnant or nursing a child may not take part in this study. You should not breastfeed while receiving nivolumab and for up to 18 weeks after the last dose of nivolumab. If you become pregnant, there may be risks to you, the embryo, or fetus. These risks are not yet known. While laboratory or animal studies have been conducted to determine possible risks, the results do not necessarily show what will happen when the drug is used in humans. No studies have been conducted to determine if nivolumab causes damage to genetic material (DNA). Because nivolumab is an antibody, the risk of damage to DNA is believed to be low. Laboratory and animal studies have not been conducted using nivolumab to determine if nivolumab may cause cancer. One study in monkeys has been conducted to evaluate the effects of nivolumab on pregnancy. The preliminary findings revealed an increase in late stage pregnancy loss as well as deaths in premature infants. These animal study findings suggest a potential risk to human pregnancy if there is continued treatment with nivolumab during pregnancy. The use of nivolumab in pregnant women has not been formally studied in clinical studies. One case has been identified of a nivolumab treated male patient with a female partner who became pregnant. The pregnancy was uneventful and at birth, the infant was slightly underweight.

If you are a woman of childbearing ability, you and the study doctor must agree on a method of birth control to use throughout the study. You must use an adequate method to avoid pregnancy while you are on the study and for up to 5 months after the last dose of nivolumab. If you think that you have

Document Approved On: 2/26/2018

gotten pregnant during the study, you must tell the study doctor immediately. Pregnant women will be taken out of the study.

**If you are a man:** the effect of the study drug on sperm is not known. To protect against possible side effects, if you are a man you should not get a sexual partner pregnant while taking nivolumab and for up to 7 months after the last dose. You and the study doctor should agree on a method of birth control to use throughout the study.

# **Requirements for Pregnancy Testing**

If you are a woman of childbearing potential, you will have a pregnancy test within 24 hours of your first dose of study medication, and then every 4 weeks during the course of this study and during your follow up visits. Pregnancy will be determined on basis of a blood or urine sample.

#### **Occurrence of Pregnancy or Suspected Pregnancy**

If you become pregnant, suspect pregnancy or if you missed your period or it is late, or if you have a change in your usual menstrual cycle (e.g., heavier bleeding during your period or bleeding between periods), you should immediately contact your study doctor.

#### **Discontinuation from the Study**

Should you become pregnant during this study, you will immediately have the study medication permanently discontinued and be referred for obstetric care. You will continue to be followed for any side effects or potential benefits of the study treatment, provided it is safe for you and your unborn baby to do so. Your doctor will discuss this with you, as well as options for additional appropriate care for your cancer. The sponsor has not set aside any funds to pay for any aspects of obstetric, child or related care and does not plan to pay for them.

#### **Pregnancy Reporting**

In case of a pregnancy, your pregnancy and its outcome will be reported to the investigator and to Bristol-Myers Squibb

#### Information for Men with Partners of Childbearing Potential

Most study drugs do not pose a risk to a woman who becomes pregnant while her male partner is a study subject. However, you are asked to inform your study doctor if your partner becomes pregnant while you are enrolled in this clinical trial, and you and your partner will be asked to provide information about the pregnancy outcome. The sponsor has not set aside any funds to pay for any aspects of obstetric, child or related care and does not plan to pay for them.

You should immediately contact your study doctor if there is a change in your method to avoid pregnancy or if you start any prescription drug or other medication (including over-the-counter drugs and herbal supplements) not prescribed by the study doctor.

If you will be taking the study drug home, keep it out of the reach of children or anyone else who may not be able to read or understand the label. Do not let anyone else take the study drug besides you.

It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this

study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

#### **Radiation Risks**

You will be exposed to radiation from CT scans. These procedures are necessary for your medical care and will occur even if you do not participate in this study. The radiation dose estimate that you will receive is equal to or less than the radiation exposure allowed to be received by a radiation worker for 3 years. The principal risk associated with a radiation dose is the possibility of developing a radiation-induced cancer later in life. Although the risk from radiation is cumulative it is not expected to adversely affect your condition or treatment. The Emory University Radiation Safety Committee has reviewed and approved the use of radiation in this research study.

### Will I benefit directly from the study?

This study is not designed to benefit you directly. Your lung cancer may improve while you are in this study but it may not, and it may even get worse. This study is designed to learn more about how nivolumab activates T cells in your immune system in the blood and in your tumor. The study results may be used to help others in the future.

#### Will I be compensated for my time and effort?

You will not be offered compensation for being in this study.

#### What are my other options?

If you decide not to enter this study, there is care available to you outside of this research study. You can still get nivolumab as standard therapy outside of this clinical trial. You may also be a candidate for other types of treatment that activate the immune system or other chemotherapy options. You may also decide that you do not want to take any treatment for your lung cancer and just treat symptoms as they develop. The study doctor will discuss these with you. You do not have to be in this study to be treated for lung cancer.

Taking part in this study, however, may make you unable to participate in some other research studies, if they exclude people who have taken certain treatments. You should discuss this with the researchers if you have concerns. You may wish to research other study options at websites like clinicaltrials.gov and ResearchMatch.org.

### How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

Study records can be opened by court order. They also may be provided in response to a subpoena or a request for the production of documents.

#### **Storing and Sharing your Information**

Your samples, genomic data and health information will be stored and shared with other researchers. The samples and information will be available for any research question, such as research to understand what causes certain diseases (for example heart disease, cancer, or psychiatric

disorders), development of new scientific methods, or the study of where different groups of people may have come from.

#### **Medical Record**

If you have been an Emory and Grady Health System patient before, then you already have an Emory and Grady Health System medical record. If you have never been an Emory and Grady Health System patient, you do not have one. An Emory and Grady Health System medical record will be made for you if an Emory and Grady Health System provider or facility gives you any services or procedures for this study.

Copies of the consent form/HIPAA authorization that you sign will be put in any Emory Healthcare medical record you have now or any time during the study.

Emory and Grady Health System may create study information about you that can help with your care. For example, the results of study tests or procedures. These study results will be put in your Emory and Grady Health System medical record. Anyone who has access to your medical records will be able to have access to all the study information placed there. The confidentiality of the study information in your medical record will be protected by laws like the HIPAA privacy rule. State and federal laws may not protect the research information from disclosure.

The results of some study tests and procedures will be used only for research purposes and will *not* be placed in your medical record. For this study, those items include any results from the immunological testing done on your blood or tumor in our research lab.

Tests and procedures done at non-Emory and Grady Health System places may not become part of your Emory and Grady Health System medical record. Also, if you decide to be in this study, it is up to you to let your other health providers know.

#### In Case of Injury

If you get ill or injured from being in the study, Emory and Grady Health System will help you get medical treatment. Emory and Grady Health System and the sponsor have not, however, set aside any money to pay you or to pay for this medical treatment. The only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory and Grady Health System or sponsor employee. "Negligence" is the failure to follow a standard duty of care.

If you become ill or injured from being in this study, your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurer does not pay, then you will have to pay these costs.

If you believe you have become ill or injured from this research, you should contact Dr. Rathi Pillai at telephone number 404-778-1900. You should also let any health care provider who treats you know that you are in a research study.

#### **Costs**

The study sponsor will pay for your study required lung biopsies and biomarker blood tests.

You will have to pay for the items or services for which the study sponsor does not pay. The sponsor will not pay for your regular medical care. If you have insurance, Emory and Grady Health System will

submit claims to your insurance for items and services that the sponsor does not cover. Emory and Grady Health System will send in only those claims for items and services that it reasonably believes your insurance will pay and that the sponsor has not paid.

The actual amount that you have to pay depends on whether or not you have health insurance and whether or not that insurance will pay for any research study costs. Generally, insurance companies will not pay for items and services that are required just for a research study. Some insurance companies will not pay for regular medical treatment or treatment for complications if you are in a study. How much you will have to pay for any co-payments, deductibles or co-insurance depends on your plan. Emory and Grady Health System and the sponsor will not pay for these costs.

It is a good idea to contact your insurance provider and tell them you want to be in this research study. Ask them what they will pay for and what they will not pay for. You can also ask the study team for help in figuring out what you will have to pay.

If you do not have insurance, Emory and Grady Health System will review your case as part of its program for low-income patient care. The standard policies of that program will apply. The program will figure out if you have to pay any costs for taking part in the study and what those costs will be.

#### Withdrawal from the Study

You have the right to leave a study at any time without penalty.

For your safety, however, you should consider the study doctor's advice about how to go off the study treatment. If you leave the study before the final planned study visit, the researchers may ask you to have some of the final steps done.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

#### Authorization to Use and Disclose Protected Health Information

The privacy of your health information is important to us. We call your health information that identifies you, your "protected health information" or "PHI." To protect your PHI, we will follow federal and state privacy laws, including the Health Insurance Portability and Accountability Act and regulations (HIPAA). We refer to all of these laws as the "Privacy Rules." Here we let you know how we will use and disclose your PHI for the main study and for any optional studies in which you may choose to participate.

#### **Main Study**

#### PHI that Will be Used/Disclosed:

The PHI that we will use or share for the main research study includes:

- Medical information about you including your medical history and present/past medications.
- Results of exams, procedures and tests you have before and during the study.

Laboratory test results.

# Purposes for Which Your PHI Will be Used/Disclosed:

We will use and share your PHI for the conduct and oversight of the research study. We will use and share your PHI to provide you with study related treatment and for payment for such treatment. We will also use and share your PHI to conduct normal business operations. We may share your PHI with other people and places that help us conduct or carry out the study, such as laboratories, data management centers, data monitors, contract research organizations, Institutional Review Boards (IRBs) and other study sites. If you leave the study, we may use your PHI to determine your health, vital status or contact information.

#### Use and Disclosure of Your Information That is Required by Law:

We will use and disclose your PHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults. We will also comply with legal requests or orders that require us to disclose your PHI. These include subpoenas or court orders.

# Authorization to Use PHI is Required to Participate:

By signing this form, you give us permission to use and share your PHI as described in this document. You do not have to sign this form to authorize the use and disclosure of your PHI. If you do not sign this form, then you may not participate in the research study or receive research-related treatment. You may still receive non-research related treatment.

# People Who will Use/Disclose Your PHI:

The following people and groups will use and disclose your PHI in connection with the research study:

- The Principal Investigator and the research staff will use and disclose your PHI to conduct the study and give you study related treatment.
- Emory and Grady Health System may use and disclose your PHI to run normal business operations.
- The Principal Investigator and research staff will share your PHI with other people and groups to help conduct the study or to provide oversight for the study.
- Emory University is the Sponsor of the study. The Sponsor may use and disclose your PHI to make sure the research is done correctly and to collect and analyze the results of the research. The Sponsor may disclose your PHI to other people and groups like study monitors to help conduct the study or to provide oversight for the study.
- Bristol Myers Squibb is a pharmaceutical company supporting this study. Your PHI may be shared with this company to help conduct the study.
- The following people and groups will use your PHI to make sure the research is done correctly and safely:
  - Emory and Grady Health System offices that are part of the Human Research Participant Protection Program and those that are involved in study administration and billing. These include the Emory IRB, the Grady Research Oversight Committee, the Emory Research and Healthcare Compliance Offices, and the Emory Office for Clinical Research.

Study No.: CA209-461

- Government agencies that regulate the research including: Food and Drug Administration
- Public health agencies.
- o Research monitors and reviewer.
- Accreditation agencies.
- Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens, your PHI may be shared with that new institution and their oversight offices. PHI will be shared securely and under a legal agreement to ensure it continues to be used under the terms of this consent and HIPAA authorization.

# Optional Study/Storage of Data/Specimens for Future Research

# PHI That Will be Used/Disclosed for Optional Study:

The PHI that we will use and/or disclose (share) for the optional research study includes:

- Medical information about you including your medical history and present/past medications.
- Results of exams, procedures and tests you have before and during the study.
- Laboratory test results.

# Purposes for which your PHI will be Used/Disclosed for Optional Study:

We will use and disclose your PHI for the conduct and oversight of the optional research study, including the administration and payment of any costs relating to subject injury.

# Authorization for This Use of PHI is Required to Participate in Optional Study, but Not in Main Study:

You do not have to authorize the use and disclosure of your PHI. If you do not authorize the use and disclosure of your PHI for the optional study, then you may not participate in the optional research study. You can still be in the main research study even if you don't participate in the optional study.

# People Who Will Use/Disclose Your PHI for Optional Study:

The following people and groups will use and disclose your PHI in connection with the optional research study:

 The same people and groups who will use and disclose your PHI for the Main Study will also do so in connection with the optional research study/storage of PHI for future research.

#### **Expiration of Your Authorization**

Your PHI will be used until this research study ends.

#### **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your information. If you want to do this, you must contact the study team in writing at:

Dr. Rathi Pillai Winship Cancer Institute of Emory University

Winship 3286-16/CA209-461 02/16/2018 PI: Rathi Pillai, MD 

Version Date:

Document Approved On: 2/26/2018

1365-C Clifton Road, NE Atlanta, GA 30322

At that point, the researchers would not collect any more of your PHI. But they may use or disclose the information you already gave them so they can follow the law, protect your safety, or make sure that the study was done properly and the data is correct.

#### Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them. The Sponsor, and people and companies working with the Sponsor on this study are not covered by the Privacy Rules. They will only use and disclose your information as described in this Consent and Authorization.

To maintain the integrity of this research study, you generally will not have access to your PHI related to this research until the study is complete. When the study ends, and at your request, you generally will have access to your PHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. If it is necessary for your health care, your health information will be provided to your doctor.

We may remove identifying information from your PHI. Once we do this, the remaining information will not be subject to the Privacy Rules. Information without identifiers may be used or disclosed with other people or organizations for purposes besides this study.

#### **Contact Information**

Contact Rathi Pillai, MD at (404) 778-1900:

- if you have any questions about this study or your part in it,
- if you feel you have had a research-related injury or a bad reaction to the study drug, or
- if you have questions, concerns or complaints about the research

Contact the Emory Institutional Review Board at 404-712-0720 or 877-503-9797 or irb@emory.edu:

- if you have guestions about your rights as a research participant.
- if you have guestions, concerns or complaints about the research.
- You may also let the IRB know about your experience as a research participant through our Research Participant Survey at <a href="http://www.surveymonkey.com/s/6ZDMW75">http://www.surveymonkey.com/s/6ZDMW75</a>.

If you are a patient receiving care from the Grady Health System and have a questions about your rights, you may contact the Office of Research Administration at research@gmh.edu.


Study No.: CA209-461

Document Approved On: 2/26/2018

# **Consent and Authorization**

# **Consent and HIPAA Authorization for Optional Study/Studies:** Please initial below if you opt to participate in and authorize use and disclosure of your PHI in the optional study/studies previously described: [OPTIONAL Second Biopsy] Initials TO BE FILLED OUT BY SUBJECT ONLY Please print your name, sign, and date below if you agree to be in the main study. By signing this consent and authorization form, you will not give up any of your legal rights. We will give you a copy of the signed form to keep. **Printed Name of Subject** \_\_\_ am / pm Signature of Subject Time (please circle) Date (18 or older and able to consent)

# TO BE FILLED OUT BY STUDY TEAM ONLY

Name of Person Conducting Informed Consent Discussion am / pm Signature of Person Conducting Date Time (please circle) Informed Consent Discussion

 Version Date:

IRB Form 04152016